CLINICAL TRIAL: NCT05148546
Title: Prospective, Randomized, Neoadjuvant Phase II Study With Combination Immuno-oncology in Primary Clear Cell Renal Cancer at Risk for Recurrence or Distant Metastases (NESCIO-trial)
Brief Title: Neoadjuvant Study With Combination Immuno-oncology for Primary Clear Cell Renal Cell Cancer
Acronym: NESCIO
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M21NSC; CA209-6DJ (Other: BMS); 2021-002360-51 (EudraCT Number)
Record Dates: First submitted 2021-11-25; First posted 2021-12-08 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Renal Cell Carcinoma
Keywords: Resectable renal cell carcinoma; Checkpoint inhibition; Immunotherapy; PD-1 inhibitor; CTLA-4 inhibitor; LAG-3 inhibitor; Nivolumab; Ipilimumab; Relatlimab; Neoadjuvant; NESCIO; M21NSC; Checkpoint blockade
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: Open-label three-arm randomized phase II trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- A: Neoadjuvant nivolumab (Experimental): Neoadjuvant 2 cycles of nivolumab 360mg every 3 weeks
  Interventions: Drug: Neoadjuvant nivolumab
- B: Neoadjuvant nivolumab + ipilimumab (Experimental): Neoadjuvant 2 cycles of nivolumab 3 mg/kg + ipilimumab 1 mg/kg every 3 weeks
  Interventions: Drug: Neoadjuvant nivolumab; Drug: Neoadjuvant ipilimumab
- C: Neoadjuvant nivolumab + relatlimab (Experimental): Neoadjuvant 2 cycles of nivolumab 360mg + relatlimab 360mg every 3 weeks
  Interventions: Drug: Neoadjuvant nivolumab; Drug: Neoadjuvant relatlimab

INTERVENTIONS:
Drug: Neoadjuvant nivolumab — Patients will receive 2 cycles of nivolumab 360mg (arm A and C) or 3mg/kg (arm B) every 3 weeks followed by a nephrectomy.
  Other Names: Opdivo
Drug: Neoadjuvant ipilimumab — Patients will receive 2 cycles of ipilimumab 1mg/kg every 3 weeks followed by a nephrectomy.
  Other Names: Yervoy
  Arms: B: Neoadjuvant nivolumab + ipilimumab
Drug: Neoadjuvant relatlimab — Patients will receive 2 cycles of relatlimab 360mg every 3 weeks followed by a nephrectomy.
  Arms: C: Neoadjuvant nivolumab + relatlimab

SUMMARY:
The NESCIO-trial is a multicenter, randomized, open-label, three-arm phase II trial investigating different combinations of neoadjuvant immunotherapy in patients with primary, resectable, intermediate to high-risk, clear-cell renal cell carcinoma. In this trial patients will be randomized 1:1:1 to receive either 2 cycles of nivolumab 360mg every 3 weeks (arm A), 2 cycles of ipilimumab 1 mg/kg + nivolumab 3 mg/kg every 3 weeks (arm B) or 2 cycles of relatlimab 360mg + nivolumab 360mg every 3 weeks (arm C), prior to surgery at week 7.

After 42 patients (14 per arm) have been recruited, an interim analysis will be performed to evaluate the observed efficacy and toxicity within each arm and either allow for early discontinuation of the treatment or continuing recruitment for the second stage. As the primary endpoint, the pathological response (decrease in tumor) will be evaluated. If at most one pathologic response in the primary tumor is observed, the treatment arm will be closed for insufficient activity on the primary tumor. If at least 2 pathologic responses are observed, 9 additional patients will be included to a total of 23 patients per cohort. A maximum of 69 patients will be recruited for this study.

Follow up will start at week 12 with a CT-scan according to the national/center's standard. Patients will be evaluated every 3 months by physical examination and lab testing for up to two years, thereafter according to institutional guidelines up to 5 years following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18 years of age;
* World Health Organization (WHO) Performance Status 0 or 1;
* Histologically confirmed resectable clear cell RCC (measurable according to RECIST 1.1), that can be biopsied, and no history of distant metastases;
* Intermediate to high risk will be based on clinical TNM and biopsy nuclear grade. These are:

  1. cT1b-cT2a grade 4 cN0 cM0
  2. cT2b grade 3 cN0 cM0
  3. cT3 any grade cN0 cM0
  4. cT4 any grade cN0 cM0
  5. cT any cN1 (fully resectable) cM0
* No other malignancies, except adequately treated and a cancer-related life-expectancy of more than 5 years;
* Patient willing to undergo triple tumor biopsies and extra blood withdrawal during screening and in case of relapse;
* No prior immunotherapy targeting CTLA-4, PD-1 or PD-L1, or LAG-3;
* No immunosuppressive medications within 2 weeks prior start immunotherapy;
* Screening laboratory values must meet the following criteria: WBC ≥ 2.0x109/L, Neutrophils ≥1.5x109/L, Platelets ≥100 x109/L, Hemoglobin ≥5.5 mmol/L, Creatinine ≤1.5x ULN, AST ≤ 1.5 x ULN, ALT ≤ 1.5 x ULN, Bilirubin ≤1.5 X ULN, normal CK and Troponin T, normal LDH;
* Women of childbearing potential must use appropriate method(s) of contraception. They should use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug;
* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study treatment;
* Women who are not of childbearing potential (i.e., who are postmenopausal), or surgically sterile as well as azoospermic men do not require contraception;
* Patient is capable of understanding and complying with the protocol requirements and has signed the Informed Consent document.

Exclusion Criteria:

* Distantly metastasized RCC;
* Brain metastases (based on symptoms);
* Non-clear cell RCC;
* No measurable lesion according to RECIST 1.1;
* Subjects with any active autoimmune disease or a documented history of autoimmune disease, or history of syndrome that required systemic steroids or immunosuppressive medications, except for subjects with vitiligo or resolved childhood asthma/atopy;
* Prior CTLA-4 or PD-1/PD-L1 or LAG-3 targeting immunotherapy;
* Radiotherapy prior or post-surgery;
* Patients will be excluded if they test positive for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody), indicating acute or chronic infection; if treated and being at least one year free from HCV patients are allowed to participate;
* Patients will be excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS);
* Allergies and Adverse Drug Reactions (like mastocytosis);
* History of severe hypersensitivity reaction to any monoclonal antibody;
* Underlying medical conditions that, in the Investigator's opinion, will make the administration of study drug(s) hazardous or obscure the interpretation of toxicity or adverse events;
* Pregnant or nursing;
* Concurrent medical condition requiring the use of immunosuppressive medications, or immunosuppressive doses of systemic or absorbable topical corticosteroids;
* Use of other investigational drugs before study drug administration 30 days and 5 half-times before study inclusion.

Relatlimab-specific exclusion Criteria:

* Participants with history of myocarditis, regardless of etiology;
* Troponin T (TnT) > 2 × institutional ULN. Participants with TnT levels between > 1 to 2 × ULN will be permitted if a repeat levels within 24 hours are ≤ 1 ULN. If TnT levels are between >1 to 2 × ULN within 24 hours, the participant may undergo a cardiac consultation and be considered for treatment, following cardiologist recommendation. When repeat levels within 24 hours are not available, a repeat test should be conducted as soon as possible. If TnT repeat levels beyond 24 hours are < 2 × ULN, the participant may undergo a cardiac consultation and be considered for treatment, following cardiologist recommendation. Notification of the decision to enroll the participant following cardiologist recommendation has to be made to the BMS Medical Monitor or designee.
* Left ventricular ejection fraction (LVEF) assessment with documented LVEF < 50% by either transthoracic echocardiogram (TTE) or multigated acquisition (MUGA) scan (TTE preferred test) within 6 months prior to start of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2022-04-28 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Pathologic response rate | At 6 weeks
  Pathologic response rate is defined as the proportion of patients demonstrating a complete pathologic or partial pathologic response, according to central revision (pathology of NKI)

SECONDARY OUTCOMES:
Safety, measured by the frequency of immune-related adverse events leading to postponing of surgery for >2 weeks | At 8 weeks
Objective response rate | At 6 weeks
  ORR is defined as the proportion of patients demonstrating a complete or partial response according to RECIST 1.1
Recurrence Free Survival (RFS) | Up to 5 years after start of treatment
  RFS is defined as the time from randomization to recurrence or death from any cause, whichever occurs first. Subjects last known to be alive, who have not experience recurrence, will be censored.
Event-free Survival (EFS) | Up to 5 years after start of treatment
  EFS is defined as the time from randomization to recurrence, distant metastasis, or death from any cause, whichever occurs first. Subjects who are event-free at the end of follow-up will be censored.
Rate of distant metastases | Up to 5 years after start of treatment
  The proportion of patients starting treatment who experience distant metastases during follow-up.
Rate of local recurrences | Up to 5 years after start of treatment
  The proportion of patients starting treatment who experience a local recurrence during follow-up.
Surgical morbidity following neoadjuvant immunotherapy | Up to 1 year after start of treatment
  Surgical complication rates according to Clavien-Dindo classification
Description of associations of TMB, fs/INDELs, HERVE-E, RNA tumor/immune signatures, and surface marker expression with tumor immune infiltrates and response | Up to 5 years after start of treatment
Cell free methylated DNA profiles following neoadjuvant immunotherapy between baseline and surgery | At 6 weeks
Collection of fresh tumor tissue for investigating TIL, scRNA and TCRseq | At 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John Haanen, Prof, Principal Investigator — Medical oncologist/researcher; Axel Bex, Prof, Principal Investigator — Urologist/researcher
Locations (2):
- Netherlands Cancer Institute, Amsterdam, North Holland, Netherlands
- Royal Free London NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No